CLINICAL TRIAL: NCT02788487
Title: A Randomized Cross-over Study of Tongue Retaining Device and Continuous Positive Airway Pressure for Treatment of Obstructive Sleep Apnea
Brief Title: Randomized Cross-over TRD and CPAP for OSA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mahidol University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: R015932011
Record Dates: First submitted 2016-05-27; First posted 2016-06-02 (Estimated); Last update posted 2016-06-02 (Estimated); Status verified 2016-05

CONDITIONS: Obstructive Sleep Apnea
MeSH Terms: conditions — Sleep Apnea, Obstructive | interventions — Continuous Positive Airway Pressure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- CPAP1 use and TRD 2use (Active Comparator): Wash-in period 1 week and Continuous positive airway pressure (CPAP) is used for 3 weeks then wash-out 1 week and Tongue retaining device (TRD) is used for another 3 weeks
  Interventions: Device: Tongue retaining device; Device: CPAP
- TRD1 use and CPAP2 use (Experimental): Wash-in period 1 week and Tongue retaining device (TRD) is used for 3 weeks then Wash-out period 1 week and Continuous positive airway pressure (CPAP) is used for another 3 weeks
  Interventions: Device: Tongue retaining device; Device: CPAP

INTERVENTIONS:
Device: Tongue retaining device — Tongue retaining device is used for 3 weeks
Device: CPAP — CPAP is used for 3 weeks
  Other Names: Continuous positive airway pressure

SUMMARY:
The objectives of this study is to compare short-term outcomes of CPAP and TRD in the treatment of obstructive sleep apnea. Study design is a randomized cross-over trial during 3-weeks period of each treatment in 36 patients. Primary outcomes are quality of life, degree of sleepiness, and severity of OSA determined by FOSQ ESS, and AHI or RDI, respectively.

DETAILED DESCRIPTION:
The objectives of this study is to compare short-term outcomes of CPAP and TRD in the treatment of obstructive sleep apnea. Study design is a randomized cross-over trial during 3-weeks period of each treatment in 36 patients. Primary outcomes are quality of life, degree of sleepiness, and severity of OSA determined by FOSQ ESS, and AHI or RDI, respectively. Wash-in period 1 week and Wash-out periods 1 week are required before start each treatment.

ELIGIBILITY:
Inclusion Criteria:

1. OSA patients aged over 18 years old at Siriraj hospital
2. Apnea-hypopnea index (AHI) 5 - 30 events/ h or AHI > 30 events/h but lowest Oxygen saturation > 70%
3. Positive consented form

Exclusion Criteria:

1. Patients with severe periodontal diseases
2. Patients with unstable medical problems i.e. poorly controlled cardiovascular diseases, cancers, cerebrovascular diseases, epilepsy, dementia, etc.
3. total sleep time less than 2 hour during previous sleep study
4. Patients who could not tolerate the side effects of CPAP or TRD
5. Patients who could not follow-up until finishing the protocol or withdraw themselves from the study for any reasons.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2016-01; Primary Completion 2016-12 (Estimated); Study Completion 2017-05 (Estimated)

PRIMARY OUTCOMES:
apnea-hypopnea index (AHI) | 3 weeks

SECONDARY OUTCOMES:
Functional outcomes of sleep questionnaire (FOSQ ) score | 3 weeks
Epworth sleepiness score (ESS) scores | 3 weeks
lowest oxygen saturation during sleep test at home | 3 weeks
side effects questionnaire | 3 weeks
satisfaction and preference of device questionnaire | 3 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Anuch - Durongphan, MD, Principal Investigator — Siriraj Hospital
Locations (1):
- Siriraj Hospital, Bangkoknoi, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Banhiran W, Durongphan A, Keskool P, Chongkolwatana C, Metheetrairut C. Randomized crossover study of tongue-retaining device and positive airway pressure for obstructive sleep apnea. Sleep Breath. 2020 Sep;24(3):1011-1018. doi: 10.1007/s11325-019-01942-z. Epub 2019 Nov 21. PMID 31754961